CLINICAL TRIAL: NCT02629510
Title: A Randomized Controlled Trial Evaluating the Efficacy of Tachosil® for Prevention of Hemorrhage After Loop Electrosurgical Excisional Procedure (LEEP) in Patients With Cervical Intraepithelial Neoplasia or Cervical Cancer
Brief Title: The Efficacy of Tachosil® for Prevention of Hemorrhage After Loop Electrosurgical Excisional Procedure (LEEP)
Acronym: TACO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jeong-Yeol Park, professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: TACO_1234
Record Dates: First submitted 2015-12-07; First posted 2015-12-14 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms | interventions — TachoSil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tachosil (Experimental): The group composed of patients whose surgical margin of cervix will be treated with Tachosil® after a loop electrosurgical excisional procedure (LEEP)
  Interventions: Drug: Tachosil
- No Tachosil (No Intervention): The group composed of patients whose surgical margin of cervix will NOT be treated with Tachosil® after a loop electrosurgical excisional procedure (LEEP)

INTERVENTIONS:
Drug: Tachosil
  Arms: Tachosil

SUMMARY:
This study is aimed at identifying the efficacy of Tachosil® for prevention of hemorrhage in patients with cervical intraepithelial neoplasia or cervical cancer after undergoing a loop electrosurgical excisional procedure (LEEP).

1. Primary endpoint:

   Bleeding period within two weeks after surgery Frequency of additional treatment due to bleeding within two weeks after surgery
2. Secondary endpoint:

Amount of bleeding within two weeks after surgery Infection frequency at external genitals, vagina and cervix within two weeks after surgery Change in life quality after surgery

DETAILED DESCRIPTION:
A loop electrosurgical excisional procedure(LEEP) is a medical technology which is very commonly used in order to treat cervical intraepithelial neoplasia and cervical cancer stage FIGO IA1, as well as diagnose the disease. Though a loop electrosurgical excisional procedure of cervix is an effective and safe procedure, it may cause discomfort due to bleeding after surgery, and there are many cases in which additional treatment shall be implemented in order to control hemorrhage.

Up to now, a number of investigators have made efforts to reduce frequency of bleeding and additional hemostasis treatment after loop electrosurgical excisional procedure of cervix. Among the methods that have been studied so far, there are methods in which albothyl solution, Monsel's solution, Tranexamic acid, Amino-Cerve, or Fibrin glue are applied to the surgical margin of cervix, of which the bleeding has been stopped by using the electrocautery method. However, none of them has been recognized to be effective in reducing the frequency of bleeding and additional hemostasis treatment after loop electrosurgical excisional procedure of cervix. Accordingly, it is required to carry out researches to find new methods.

Tachosil, as an absorbable hemostatic surgical patch, is composed of collagen matrix on which coagulation factor, human fibirinogen and human thrombin are coated. It has been proved that Tachosil is an effective and safe styptic in a digestive, hapatobiliary, pulmonary, renal surgery. Unlike the existing styptic, the surgical patch Tachosil has strong adhesion to bleeding points, plugging up bleeding holes, so that it is expected to have a great effect on prevention of bleeding on surgical margin of cervix after loop electrosurgical excisional procedure of cervix.

This study is aimed at evaluating if the application of Tachosil is effective for prevention of bleeding after a loop electrosurgical excisional procedure of cervix.

ELIGIBILITY:
Inclusion Criteria

* Over 20 years old
* Patients who have to undergo a loop electrosurgical excisional procedure as they have been diagnosed with cervical intraepithelial neoplasia or cervical cancer, including patients whose symptoms are suspicious for such diseases.
* Patients who are able to sign a informed consent, and who have signed.

Exclusion Criteria

* Patients who have experienced a treatment due to diagnosis of cervical intraepithelial neoplasia or cervical cancer
* Patients who have a disease of bleeding tendancy, or patients who have taking drugs.
* Patients with abnormal uterine bleeding or vaginal bleeding.
* Patients with active medical disease
* Patients with uncontrollable medicall disease
* Patients who are pregnant or breastfeeding
* Patients who can not participate in the clinical study due to legal restrictions

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Estimated)
Dates: Start 2015-01; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Bleeding period after surgery in days | two weeks

SECONDARY OUTCOMES:
Amount of bleeding after surgery | two weeks
  evaluated by using the Pictorial Bleeding Assessment Chart
Infection frequency at external genitals, vagina and cervix after surgery | two weeks
  infection frequency is counted by record of treatment for infectious disease for two weeks after surgery and pelvic examination when the patients is visiting the hospital on the second week after surgery
Change in life quality after surgery | 4 weeks prior to, during the period between 14 and 21 days after, and 6 weeks after, respectively
  evaluated three times by using the Medical Outcomes Study Short-Form-36 (SF-36)
Amount of vaginal discharge | two weeks
  measuring the amount of vaginal discharge on the day when there is no vaginal bleeding by using a visual analogue scale, the amount will be scored on a scale ranging from 0 to 5 the day when there is no discharge at all is defined as 0, and the day when the patient has experienced the most amount of discharge is defined as 5 on the five-point scale
Frequency of additional treatment due to bleeding after surgery | two weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim J, Park JY. Hemostatic Efficacy of TachoSil in Loop Electrosurgical Excisional Procedure: A Prospective Randomized Controlled Study. J Low Genit Tract Dis. 2025 Apr 1;29(2):123-130. doi: 10.1097/LGT.0000000000000867. Epub 2025 Jan 22. PMID 39842025